CLINICAL TRIAL: NCT00060008
Title: Novel Imaging Modalities For Plexiform Neurofibromas
Brief Title: Fludeoxyglucose F 18 Positron Emission Tomography and Magnetic Resonance Perfusion Imaging in Patients With Neurofibromatosis 1 and Plexiform Neurofibroma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was closed early due to poor accrual.
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2001-8-2543; CHP-724 (Other: Children's Hospital of Philadelphia); CDR0000299006
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Neurofibromatosis Type 1; Precancerous Condition
Keywords: neurofibromatosis type 1; plexiform neurofibroma
MeSH Terms: conditions — Neurofibromatosis 1; Precancerous Conditions; Neurofibroma, Plexiform | interventions — Fluorodeoxyglucose F18; Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18FDG-PET scan and MR perfusion (Experimental): Subjects will undergo MRI for quantitative (2D and 3D) evaluation of plexiform neurofibroma size, MR perfusion scan, and fludeoxyglucose (18FDG) PET scan at the time of study entry. Subjects who are treated for plexiform neurofibroma will undergo another 18FDG PET scan after one year of study entry.
  Interventions: Radiation: fludeoxyglucose F 18; Radiation: gadopentetate dimeglumine

INTERVENTIONS:
Radiation: fludeoxyglucose F 18
Radiation: gadopentetate dimeglumine

SUMMARY:
RATIONALE: New imaging procedures such as fludeoxyglucose F 18 positron emission tomography (FDG-PET) and magnetic resonance (MR) perfusion imaging may improve the ability to detect disease progression, help doctors predict a patient's response to treatment, and help plan the most effective treatment.

PURPOSE: This diagnostic trial is studying how well FDG-PET and MR perfusion imaging work in finding disease progression and determining response to treatment in patients with neurofibromatosis 1 and plexiform neurofibroma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether fludeoxyglucose F 18 positron emission tomography (FDG-PET) and MR perfusion studies can predict plexiform neurofibroma growth rates in patients with neurofibromatosis 1.
* Determine whether FDG-PET and MR perfusion studies can predict the likelihood of response in patients who are undergoing investigational treatment for plexiform neurofibromas.
* Identify neuroimaging characteristics that distinguish patients who have responded to therapy from those who have not after completion of treatment.

OUTLINE:

* Stratum 1: Patients undergo MR perfusion scan with gadopentetate dimeglumine and fludeoxyglucose F 18 positron emission tomography (FDG-PET) at baseline and quantitative MRI evaluation at baseline and 1 year.
* Stratum 2: Patients undergo quantitative MRI, MR perfusion scan with gadopentetate dimeglumine, and FDG-PET at baseline and 1 year.

PROJECTED ACCRUAL: A total of 48 patients (32 for stratum 1 and 16 for stratum 2) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Stratum 1:

  * Diagnosis of neurofibromatosis 1 (NF1) and plexiform neurofibromas
  * At high risk for progression, as defined by any of the following:

    * Anatomic location such that progression carries a high risk of impairment of function, pain, or disfigurement (e.g., neck/mediastinum, paraspinal nerve roots, orbit, and face)
    * Tumors that the patient, family, or caregiver believes have increased in size within the past year, but appear stable by standard clinical or radiographic measures
  * No plexiform neurofibromas that are small, cause no pain or functional impairment, or are not likely to cause pain or functional impairment over the succeeding 12 months
* Stratum 2:

  * Diagnosis of NF1 and progressive plexiform neurofibromas

    * Neurofibroma progression documented by increase in lesion size on MRI
  * Currently being enrolled on a clinical therapeutic trial at Children's Hospital of Philadelphia

PATIENT CHARACTERISTICS:

Age

* 25 and under

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Stratum 1:

  * No prior or concurrent chemotherapy
  * No concurrent enrollment on a chemotherapy clinical trial
* Stratum 2:

  * At least 4 weeks since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 6 weeks since prior radiotherapy (stratum 2)

Surgery

* Prior surgery for progressive plexiform neurofibroma allowed if incompletely resected and measurable disease remains (stratum 2)

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2002-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fisher, MD, Study Chair — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- 18FDG-PET Scan and MR Perfusion: Subjects will undergo MRI for quantitative (2D and 3D) evaluation of plexiform neurofibroma size, MR perfusion scan, and fludeoxyglucose (18FDG) PET scan at the time of study entry. Subjects who are treated for plexiform neurofibroma will undergo another 18FDG PET scan after one year of study entry.
  fludeoxyglucose F 18
  gadopentetate dimeglumine
Period: Overall Study
Arm/Group | 18FDG-PET Scan and MR Perfusion
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 18FDG-PET Scan and MR Perfusion
Number analyzed (Participants) | 18
Age, Customized [Mean (Full Range); unit: years] | 14.4 [6 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Tumor Progression as Measured by Tumor Area and Volume at 1 Year.
Description: We correlated SUVmax and change in tumor volume over the subsequent year
Time Frame: One year
Measure: Median (Full Range); unit: percentage of change
Units Other Than Participants: tumors
Groups:
- SUVmax < 2; SUVmax >2: Subjects underwent MRI for quantitative (3D) evaluation of plexiform neurofibroma size and fludeoxyglucose (18FDG) PET scan at the time of study entry.
Arm/Group | SUVmax < 2 | SUVmax >2
Number analyzed (Participants) | 11 | 4
Number analyzed (tumors) | 15 | 4
percentage of change | 4 [-0.6 to 63] | 27 [16 to 32]
Statistical Analysis 1: Comparison: SUVmax < 2 vs SUVmax >2; Test type: Superiority or Other; p = 0.016, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Description: Adverse Events were not collected for this study.
Arm/Group | 18FDG-PET Scan and MR Perfusion
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The sample size was modest. It is possible that with increased sample size, if the correlation estimate holds, it will become statistically significant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No